CLINICAL TRIAL: NCT05017792
Title: Evaluation of Clinical and Antibody Response to Covid-19 Vaccination Strategy in TBRI, Egypt
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samia Hassan El-Shishtawy (Other)
Responsible Party: Sponsor-Investigator, Samia Hassan El-Shishtawy, assistant professor, Theodor Bilharz Research Institute
Organization: Theodor Bilharz Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 00022021
Record Dates: First submitted 2021-08-23; First posted 2021-08-24 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 5 blood samples will be taken: Each one is 5 cm as following
  1- Before vaccination:
  To detect:
  * COVID-19 IgG/IgM Rapid Test
  * COVID-19 IgG/IgM by quantitative method(ELISA).
  * D-dimer
  * COVID-19 IgM detection
  * COVID-19 IgG detection D-dimer Measuring D-dimer 3-Before the second dose: To detect IgG and IgM To detect the level of Covid-19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
    4-After 3 months from the second dose: To detect the level ofCovid-19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
    5-After 6 months from the second dose: To detect the level ofCovid 19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 1- Before vaccination: (Other): To detect:
  * COVID-19 IgG/IgM Rapid Test
  * COVID-19 IgG/IgM by quantitative method(ELISA).
  * D-dimer
  Interventions: Biological: Astrazenica vaccine
- 2-7 days after the first dose (Other): Measuring D-dimer
  Interventions: Biological: Astrazenica vaccine
- 3-Before the second dose: (Other): To detect IgG and IgM To detect the level of Covid-19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
  Interventions: Biological: Astrazenica vaccine
- 4-After 3 months from the second dose: (Other): To detect the level ofCovid-19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
  Interventions: Biological: Astrazenica vaccine
- 5-After 6 months from the second dose: (Other): To detect the level ofCovid 19 Ig G antibodies titer in the blood, Quantitative Ig G titer should be measured. To detect the response of the immune system to the vaccine.
  Interventions: Biological: Astrazenica vaccine

INTERVENTIONS:
Biological: Astrazenica vaccine — COVID-19 vaccines should be administered by intramuscular (IM) injection, preferably into the deltoid muscle of the upper arm. Individuals who have minimal muscle mass in the deltoid area of the upper arm, or a particular reason to avoid immunization in the deltoid muscle, can be given their vaccine in the vastuslateralis muscle in the thigh if necessary.

SUMMARY:
Evaluation of the efficacy of the AstrazenicaCovid 19 vaccine to develop IgG antibody and its level based on th12 weeks program. Also to follow the changes of markers of coagulation (D-dimer) after vaccination compared to the basic level. A cardiology consultant will follow D-Dimer results to be managed properly if there is a need. As it is expected to receive Sinopharm vaccine there will be comparison between results of the two types of vaccine. To our knowledge this will be the first study done on Egyptian population.

DETAILED DESCRIPTION:
SARS-CoV-2 has been in the human population for more than a year now, causing severe disease in some and resulting in a pandemic that continues to put severe strain on economies and healthcare infrastructures worldwide. Vaccination is considered as one of the greatest successes in medical history. Based on prior experience with the development of SARS-CoV vaccines, all COVID-19 vaccines must be subjected to the tests for protective effects and harmful risks derived from antibody-dependent enhancement that may contribute to augmented infectivity and/or eosinophilic infiltration. The SARS-CoV-2 vaccine is now being developed urgently in several different ways.

In the UK, the first three vaccines have emergency use authorization, and a national rollout is in progress. Many other countries are also instigating large scale vaccination programmes. Assessment of the safety and efficacy of vaccines against the severe acute respiratory syndrome coronavirus (SARS-CoV-2) in different populations is essential .

The UK government recently decided to extend the interval between the first dose of the Pfizer BioNTech and AstraZeneca COVID-19 vaccines from 3 weeks to 12 weeks to maximise the number of people receiving the initial dose, despite the trials only providing vaccine efficacy data based on a schedule of 21 days between doses.

Many reports were raised claiming Astrazenica vaccine for the development of vascular thrombosis and studies are not finalized regarding this issue .

China is regarded as one of the world's leading countries in SARS-CoV-2 vaccine development, up to date the last inactivated vaccine international clinical (Phase III) trial was launched in the United Arab Emirates by Sinopharm China National Biotec Group (CNBG).The ability to track and trace vaccines through the vaccine supply chain down to persons vaccinated has to be enhanced.

ELIGIBILITY:
Inclusion Criteria:

* All male and female above 18 years

Exclusion Criteria:

* age below 18 years -pregnancy-
* fever
* IGM positive for covid 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — ABOVE 18 YEARS
Enrollment: 200 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
to develop IgG antibody | seven to ten days
  These antibodies indicate that you may have had COVID 19 in the recent past and have developed antibodies that may protect you from future infection. It is unknown at this point how much protectionantibodies might provide against reinfection. This group of individuals should receive the vaccine. Quantitative Ig G titer should be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Samia El-Shishtawy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No